CLINICAL TRIAL: NCT03024021
Title: The Effect of Cerebral Oxymetry in Determining Neurological Outcome in Patients Treated With Therapeutic Hypothermia
Brief Title: Cerebral Oxymetry and Neurological Outcome in Therapeutic Hypothermia
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aykut Saritas, principal investigator, Tepecik Training and Research Hospital
Other Study IDs: 29/3
Record Dates: First submitted 2016-12-21; First posted 2017-01-18 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Post-Cardiorespiratory Arrest Coma; Cardiac Arrest
Keywords: therapeutic hypothermia; targeted temperature management; neurological outcome; post-cardiac arrest syndrome
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Heart Arrest; Post-Cardiac Arrest Syndrome | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Near-infrared spectroscopy (NIRS) (INVOS®, Covidien) — As we start the targeted temperature management protocol (24 hours of hypothermia adjusted to 33-36 C and afterwards up to five days of normothermia [36.5 C]) NIRS sensor pads will be placed over the right and left frontal area. Regional cerebral oxygen values will be continuously recorded at the NIRS monitor. Tests to assess neurological outcome will be performed. Patients will be assessed in terms of neurological performance tests and regional cerebral oxygen.

SUMMARY:
This study is designed to assess the effect of cerebral oxygen saturation as an early predictor of neurological outcomes in patients undergoing therapeutic hypothermia after cardiac arrest

DETAILED DESCRIPTION:
Our study is planned as a prospective observational study. Patients undergoing therapeutic hypothermia in our intensive care unit after cardiac arrest will be enrolled. Each patient's cerebral oxygenation will be monitored with near-infrared spectroscopy (NIRS) in every 6 hours during our 24 hour lasting hypothermia period. Afterwards, patients will be monitorised in every 6 hours during the first day of hypothermia and than the mean values of daily cerebral oxygen values will be noted in the third, fourth and fifth days of nomothermia. Regional oxygen saturation (rSO2) will be noted from left and right probes. Full Outline of Unresponsiveness (FOUR) Score, Glasgow Coma Score (GCS) and cerebral performance category scale (CPC) will be noted at the beginning of therapeutic hypothermia and each day during normothermia, day 21 and the day of discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patients undergoing therapeutic hypothermia

Exclusion Criteria:

* Patients under 18 years
* Patients unsuitable for therapeutic hypothermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing therapeutic hypothermia after cardiac arrest in a tertiary intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Measure of cerebral oximetry | 8 times during the first 48 hours of hospitalization
  During the first 48 hours of hospitalization, we will collect the cerebral oximetry values in the two cerebral. hemispheres.

SECONDARY OUTCOMES:
The cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor neurological outcome according with CPC score | Participants will be followed for 8 times during the first 48 hours of hospitalization, the third day, fourth day and fifth day and the duration of hospital stay, an expected average of 2-4 weeks and a 12 month follow up will be performed
  The cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor neurological outcome according to the CPC score.
  CPC 1: Conscious and alert with normal function or only slight disability CPC 2: Conscious and alert with moderate disability CPC 3: Conscious with severe disability CPC 4: Comatose or persistent vegetative state CPC 5: death. CPC will be evaluated at the time of admission to intensive care unit and day 21.CPC score (CPC = 1 become good score - 2 and bad become CPC = 3-5).

OTHER OUTCOMES:
The cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor neurological outcome according with Four score | Participants will be followed for 8 times during the first 48 hours of hospitalization, the third day, fourth day and fifth day and the duration of hospital stay, an expected average of 2-4 weeks and a 12 month follow up will be performed
  The cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor neurological outcome according to the Fourscore (Full Outline of UnResponsiveness):It evaluates four functional categories: eye response, motor response, brainstem reflexes, and respiration pattern (including mechanical ventilation). All the four categories are scored from 0 to 4 points, with 4 representing normal, and 0 indicating no function.

CONTACTS AND LOCATIONS:
Overall Officials: Aykut Saritas, Study Director — Tepecik Research and Training Hospital; Burcu Acar Cinleti, Study Chair — suat seren research and training hospital; Ciler Zincircioglu, Study Chair — Tepecik Research and Training Hospital; İsil Kose, Study Chair — Tepecik Research and Training Hospital; Ugur Uzun, Study Chair — Tepecik Research and Training Hospital; Nimet Senoglu, Study Chair — Tepecik Research and Training Hospital
Locations (1):
- Tepecik Research and Training Hospital, Izmir, Konak, Turkey (Türkiye)

REFERENCES:
- [Background] Storm C, Leithner C, Krannich A, Wutzler A, Ploner CJ, Trenkmann L, von Rheinbarben S, Schroeder T, Luckenbach F, Nee J. Regional cerebral oxygen saturation after cardiac arrest in 60 patients--a prospective outcome study. Resuscitation. 2014 Aug;85(8):1037-41. doi: 10.1016/j.resuscitation.2014.04.021. Epub 2014 Apr 30. PMID 24795284
- [Result] Genbrugge C, Eertmans W, Meex I, Van Kerrebroeck M, Daems N, Creemers A, Jans F, Boer W, Dens J, De Deyne C. What is the value of regional cerebral saturation in post-cardiac arrest patients? A prospective observational study. Crit Care. 2016 Oct 13;20(1):327. doi: 10.1186/s13054-016-1509-9. PMID 27733184
- [Result] Nishiyama K, Ito N, Orita T, Hayashida K, Arimoto H, Beppu S, Abe M, Unoki T, Endo T, Murai A, Hatada T, Yamada N, Mizobuchi M, Himeno H, Okuchi K, Yasuda H, Mochizuki T, Shiga K, Kikuchi M, Tsujimura Y, Hatanaka T, Nagao K; J-POP Registry Investigators. Regional cerebral oxygen saturation monitoring for predicting interventional outcomes in patients following out-of-hospital cardiac arrest of presumed cardiac cause: A prospective, observational, multicentre study. Resuscitation. 2015 Nov;96:135-41. doi: 10.1016/j.resuscitation.2015.07.049. Epub 2015 Aug 17. PMID 26291387